CLINICAL TRIAL: NCT02464891
Title: An Open-label Phase 2 Study to Assess the Effect of C5aR Antagonist Therapy by CCX168 Oral Administration on ex Vivo Thrombus Formation and Disease Activity in ESRD Patients With Atypical Hemolytic Uremic Syndrome
Brief Title: Complement Inhibition in aHUS Dialysis Patients
Acronym: ACCESS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study had accomplished its goal with the 6 patients who have been enrolled.
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL006_168; 2014-004261-24 (EudraCT Number)
Record Dates: First submitted 2015-05-26; First posted 2015-06-08 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Atypical Hemolytic Uremic Syndrome
Keywords: Atypical Hemolytic Uremic Syndrome; CCX168; dialysis; C5aR antagonist
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome | interventions — avacopan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CCX168 (Experimental): Study medication will be administered as hard gelatin capsules containing 10 mg CCX168. Patients will take 30 mg CCX168, given as 3 x 10 mg capsule, twice daily for 15 days.
  Interventions: Drug: CCX168

INTERVENTIONS:
Drug: CCX168

SUMMARY:
This study evaluates the effect of CCX168, a C5aR Antagonist, Oral Administration on Ex Vivo Thrombus Formation and Disease Activity in ten patients with diagnosis of Atypical Hemolytic Uremic Syndrome with or without genetic abnormalities in the complement system or thrombomodulin, on stable chronic extracorporeal or peritoneal dialysis therapy since at least 6 months.

DETAILED DESCRIPTION:
Inherited defects that determine uncontrolled activation of the alternative complement pathway have been well documented in atypical Hemolytic Uremic Syndrome (aHUS) patients. Research in recent years has identified more than 120 different mutations, accounting for around 40%-60% of cases, in the genes encoding complement factor H (CFH), membrane cofactor protein (MCP), complement factor I (CFI), C3, complement factor B (CFB), and thrombomodulin (THBD). A therapeutic approach could be the administration of molecules that pharmacologically target complement activation, which is the primary common pathogenic mechanism in all genetic forms of aHUS. Eculizumab has been successfully used as prophylaxis of aHUS recurrences in subjects with plasma dependent or plasma resistant disease or in renal transplant recipients at high risk of recurrence due to CFH, CFI, or C3 complement gene mutations. However the drug must be administered chronically and drug spacing or discontinuance was associated with disease recurrence in the graft. The C5aR receptor antagonist CCX168 could present an appealing alternative to eculizumab for post-transplant prophylaxis of aHUS recurrences since it is orally administrable with lower cost of goods. In addition, CCX168 is theoretically associated with lower risk of infections than eculizumab since the former does not target C5b and leaves the terminal complement pathway intact.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years;
* Diagnosis of aHUS with or without identified genetic abnormalities in the complement system or thrombomodulin;
* Stable chronic extracorporeal or peritoneal dialysis therapy since at least 6 months;
* Written informed consent.

Exclusion Criteria:

* Women of childbearing potential or women who are breastfeeding;
* Shiga toxin-associated HUS or secondary forms of thrombotic microangiopathy;
* ADAMTS13 activity <10 % or circulating anti ADAMTS13 autoantibodies consistent with the diagnosis of thrombotic thrombocytopenic purpura;
* Need for specific intervention with plasma therapy and/or complement inhibitors as deemed clinically appropriate;
* Plasma therapy or treatment with complement inhibitors or antiplatelet and antithrombotic agents over the last two weeks;
* Liver function impairment (serum liver enzymes or bilirubin levels >3 x upper limit of normal);
* Neutrophil count < 2000/μL or lymphocyte count < 1000/μL;
* Infection requiring antibiotic treatment within the previous 4 weeks prior to screening;
* Participated in any clinical study of an investigational product within 30 days prior to screening or within 5 half-lives after taking the last dose;
* History or presence of any medical condition or disease which, in the opinion of the Investigator may place the subject at unacceptable risk for study participation;
* Inability to understand the potential risks and benefits of the study;
* Legal incapacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-06-04 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2017-07-13 (Actual)

PRIMARY OUTCOMES:
Ex vivo thrombogenesis. | Changes from baseline at day 2,14 (during CCX168 treatment), 16 and 21 (after treatment withdrawal).

SECONDARY OUTCOMES:
Complement component 3 serum levels. | Changes from baseline at day 2,14 (during CCX168 treatment), 16 and 21 (after treatment withdrawal).
Complement component 4 serum levels. | Changes from baseline at day 2,14 (during CCX168 treatment), 16 and 21 (after treatment withdrawal).
Complement component 5 serum levels. | Changes from baseline at day 2,14 (during CCX168 treatment), 16 and 21 (after treatment withdrawal).
Complement Factor H. | Changes from baseline at day 2,14 (during CCX168 treatment), 16 and 21 (after treatment withdrawal).
Complement component 5a. | Changes from baseline at day 2,14 (during CCX168 treatment), 16 and 21 (after treatment withdrawal).
Soluble thrombomodulin. | Changes from baseline at day 2,14 (during CCX168 treatment), 16 and 21 (after treatment withdrawal).
Fibrin split products.. | Changes from baseline at day 2,14 (during CCX168 treatment), 16 and 21 (after treatment withdrawal).
Ex vivo C5b-9 deposition on microvascular endothelial cells | At baseline.
Changes in pre-dialysis and intradialytic blood pressure. | The participants will be followed for the duration of the study up to 21 days.
Changes in heart rate. | The participants will be followed for the duration of the study up to 21 days.
Safety and tolerability parameters including serious and non serious events | The participants will be followed for the duration of the study up to 21 days.
Patient health-related quality of life as measured by administration of EQ-5D-5L questionnaire. | Changes from baseline at 14 and 21 day.
Characterization of CCX168 pharmacokinetic profile after oral administration by determining by maximum plasma concentration, time of maximum plasma concentration and area under the plasma concentration-time curve from time 0 to hour 6 | Changes from Baseline at 4,9,11 and 15 day.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Remuzzi, MD, Study Chair — IRCCS - Mario Negri Institute for Pharmacological Research/A.O. Papa Giovanni XXIII- BG
Locations (1):
- A.O. Papa Giovanni XXIII - U.O. Nefrologia e Dialisi/IRCCS IRFMN - Centro di Ricerche Cliniche per le Malattie Rare Aldo e Cele Daccò, Bergamo, Italy

REFERENCES:
- [Derived] Aiello S, Gastoldi S, Galbusera M, Ruggenenti P, Portalupi V, Rota S, Rubis N, Liguori L, Conti S, Tironi M, Gamba S, Santarsiero D, Benigni A, Remuzzi G, Noris M. C5a and C5aR1 are key drivers of microvascular platelet aggregation in clinical entities spanning from aHUS to COVID-19. Blood Adv. 2022 Jan 8;6(3):866-881. doi: 10.1182/bloodadvances.2021005246. PMID 34852172